CLINICAL TRIAL: NCT05090644
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: Program for the Introduction Into Clinical Practice of the Principles of Personalized and Preventive Medicine Based on the Isolation of Gene Polymorphism in Schizophrenia in People of the Kazakh Ethnic Group
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1203
Record Dates: First submitted 2021-09-25; First posted 2021-10-25 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia
Keywords: GWAS
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: Patients with schizophrenia
  Interventions: Genetic: DNA analysis
- Control group: Patients without schizophrenia
  Interventions: Genetic: DNA analysis

INTERVENTIONS:
Genetic: DNA analysis — GWAS

SUMMARY:
This is a GWAS study that aims to identify possible candidate genes associate to schizophrenia by exploring single nucleotide polymorphism (SNP) in a group of schizophrenia, in the Kazakh population. The investigators hypothesize that the careful phenotyping of the subject sand matching with increase the power to find SNP significantly associated with schizophrenia

DETAILED DESCRIPTION:
A genome-wide association study (GWAS) is an approach used in genetics research to associate specific genetic variations with particular diseases. The method involves scanning the genomes from many different people and looking for genetic markers that can be used to predict the presence of a disease. Once such genetic markers are identified, they can be used to understand how genes contribute to the disease and develop better prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* persons of Kazakh nationality having this ethnicity in the 3rd generation
* age from 18 to 65 years old;
* the dispensary in a psychiatric institution at the place of residence with a diagnosis of "Paranoid schizophrenia";
* the duration of the disease is at least 1 year (from the moment of taking under dispensary supervision):
* absence of severe and chronic somatic diseases;
* absence of severe and chronic neurological diseases;
* absence of comorbid drug addiction pathology;
* signed informed consent to conduct this study

Exclusion Criteria:

* persons of non-Kazakh nationality and Kazakh nationality, not confirmed until the 3rd generation
* age less than 18 years old and over 65 years old;
* those who are on dispensary registration in a psychiatric institution at the place of residence with a diagnosis not related to ICD-10 under the heading F20.0 "Paranoid schizophrenia";
* having a disease duration of less than 1 year (from the moment of taking under dispensary supervision):
* having severe and chronic somatic diseases;
* having severe and chronic neurological diseases;
* having comorbid narcological pathology;
* not signed informed consent to conduct this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Kazakh population
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
number of SNPs associated with schizophrenia | 1 year
  Using GWAS to identify candidate genes associate with schizophrenia

CONTACTS AND LOCATIONS:
Overall Officials: Kuanysh Altynbekov, PhD, Principal Investigator — Republican Scientific and Practical Center for Mental Health
Locations (1):
- Republican Scientific and Practical Center for Mental Health, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided